CLINICAL TRIAL: NCT03313453
Title: Effect of Air Cleaner on the Indoor Allergen Sensitized Allergic Rhinitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2017-0588
Record Dates: First submitted 2017-09-29; First posted 2017-10-18 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation of intervention arm and scoring of symptom and medication scire will be performed by a designated unblinded member of the study staff (i.e. a qualified person who is independent of the protocol-defined study assessments). Once prepared, active air-cleaner and mock device will be identical in appearance. The blinding of all those involved in the evaluation of the study treatment (e.g. physician/nurse as well as the subject) shall be maintained at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aircleaner group (Experimental): PuriCare (HEPA Air Cleaner) in active mode
  Interventions: Device: PuriCare (HEPA Air Cleaner)
- Control comparator (Placebo Comparator): Mock device of PuriCare in active mode
  Interventions: Device: Mock device of PuriCare

INTERVENTIONS:
Device: PuriCare (HEPA Air Cleaner) — The active comparator group is a group that uses machines that have the same functions as those on the market. In intervention group, two air-cleaners will be activated, one in the living room (covers 91 m2) and the other in the bedroom (covers 58 m2). The air cleaner will be operated continuously for 6 weeks. Inside the air cleaner, a device for measuring the quality of the indoor air is built in. It will be used to compare indoor air quality before and after air cleaner operation. In order to maintain the double-blind setting, a label for 'prohibition of opening' will be attached to the joint of the outer case, and a sticker to cover the air quality measurement display part built in the air cleaner itself will be attached.
  Arms: Aircleaner group
Device: Mock device of PuriCare — The Control group operates the air-cleaner with the same appearance as the experiment group. However, all the filters including HEPA filter will not be inserted in this group (mockup devices). Two mockup air-cleaners will be activated, one in the living room (covers 91 m2) and the other in the bedroom (covers 58 m2). The mockup devices will be operated continuously for 6 weeks. Same as active comparator group, a device for measuring the quality of the indoor air is built in the mockup air cleaner. It will be used to compare indoor air quality before and after air cleaner operation. In order to maintain the double-blind setting, a label for 'prohibition of opening' will be attached to the joint of the outer case, and a sticker to cover the air quality measurement display part built in the air cleaner itself will be attached.
  Arms: Control comparator

SUMMARY:
This study aimed to assess the impact of air cleanser on allergic rhinitis patients and indoor air quality. Air cleaners will be installed in the bedrooms and living rooms of the mite allergic rhinitis patients who aged 18-60 years.

Main parameters:

- Symptom medication score of allergic rhinitis

Supportive parameters:

* Visual analog scale of allergic rhinitis
* Quality of life score of allergic rhinitis
* Indoor air quality measurement
* Indoor allergen level measurement

DETAILED DESCRIPTION:
The most important principle in the treatment of allergic diseases is to avoid or reduce exposure to the causative antigen. Causative agents that induce allergic diseases or exacerbate symptoms are classified into indoor and outdoor allergens. House dust mites and pet's hair are typical indoor antigens. Air pollution as well as allergens are important deterioration factors, and environmental management is essential for alleviating symptoms of allergic diseases. Therefore, we are about to evaluate the impact of the air cleaner to the allergic rhinitis patients.

A total of 45 patients will be enrolled in the study and a real air cleaner and a mock-up air cleaner will be randomly installed at ratio of 1: 1 to measure rhinitis symptoms and the changes in indoor air quality after 6 weeks of operation.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 19 and 65 years of age
* Allergy specialist diagnosis of Moderate to severe persistent allergic rhinitis
* Retrospective Rhinoconjunctivitis total symptom score higher than 7
* Allergy against house dust mite: Skin prick test, with a more than 3 mm wheal, Serum specific IgE higher than 0.35 kUA/L measured by ImmunoCAP
* Who can read and write Korean
* Participants those who voluntarily agreed to this study

Exclusion Criteria:

* Allergy against seasonal allergens (tree, grass, weed pollens)
* Patients with rhinitis due to other causes (drug induced rhinitis or infectious rhinitis etc.)
* Patients with severe anatomical abnormality that may cause nasal blockage such as nasal septum deviation or nasal polyps
* Chronic systemic corticosteroids (≥ 3 months continuous use in past 12 months)
* Participants planning to move or change residence within the study period.
* Staying away from the home continuously for more than 5 days in the study period.
* Having air cleaner previously
* Having indoor smoker
* If pregnancy test is positive or pregnancy is possible during study period.
* Any other reason the participants is deemed unsuitable for participation in clinical trials

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Daily symptom score of allergic rhinitis | 6 weeks
  Daily symptom score of allergic rhinitis:
  * Rhinorrhea
  * Nasal itchiness
  * Sneezing
  * Obstruction
Daily medication score of allergic rhinitis | 6 weeks
  Daily medication score of allergic rhinitis - Intranasal steroid
  * Anti-histamine
  * Leukotriene modifier

SECONDARY OUTCOMES:
Visual analog scale of allergic rhinitis | 6 weeks
  0 to 10 score of VAS
Quality of life score of allergic rhinitis | 6 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Allergy and Immunology Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park HK, Cheng KC, Tetteh AO, Hildemann LM, Nadeau KC. Effectiveness of air purifier on health outcomes and indoor particles in homes of children with allergic diseases in Fresno, California: A pilot study. J Asthma. 2017 May;54(4):341-346. doi: 10.1080/02770903.2016.1218011. Epub 2016 Oct 10. PMID 27723364
- [Derived] Park KH, Sim DW, Lee SC, Moon S, Choe E, Shin H, Kim SR, Lee JH, Park HH, Huh D, Park JW. Effects of Air Purifiers on Patients with Allergic Rhinitis: a Multicenter, Randomized, Double-Blind, and Placebo-Controlled Study. Yonsei Med J. 2020 Aug;61(8):689-697. doi: 10.3349/ymj.2020.61.8.689. PMID 32734732